CLINICAL TRIAL: NCT06692348
Title: A Phase 1, Open-Label, Multiple-Dose Study to Investigate the Comparability of the Pharmacokinetics of Orforglipron (LY3502970) Single Capsule and Multiple Capsules in Healthy Participants
Brief Title: A Study of Orforglipron (LY3502970) to Compare a Single Capsule and Multiple Capsules in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 27228; J2A-JE-GZPM (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Orforglipron (Experimental): Participants will receive different sequences of Orforglipron doses administered as either single capsule or multiple capsules at different dose levels under either fasted or fed condition.
  Interventions: Drug: Orforglipron

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970

SUMMARY:
The main purpose of this study is to assess and compare a single capsule and multiple capsules of Orforglipron based on the amount that gets into the blood stream and how long it takes the body to get rid of it, when given to healthy participants under fasted and fed conditions. How the body handles and eliminates the study drug after meals and on an empty stomach will be measured. Information about any adverse effects experienced will be collected and the safety and tolerability of Orforglipron will also be evaluated. The study will last approximately 21 weeks, including a screening period.

ELIGIBILITY:
Inclusion Criteria:

* Have a stable body weight, that is, less than a 5% body weight change, for 1 month prior to randomization and body mass index (BMI) within the range 23.0 to 35.0 kilogram per square meter (kg/m²), inclusive
* Have safety laboratory test results within normal reference range for the population or investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have a hemoglobin A1c (HbA1c) test level greater than or equal to 6.5%
* Have an estimated glomerular filtration rate less than 30 milliliter per minute per 1.73 square meter (mL/min/1.73m²)
* Have a history of significant active or unstable major depressive disorder or other severe psychiatric disorder, for example, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder within the 2 years prior to screening
* Actively suicidal and therefore deemed to be at significant risk for suicide
* Have a known clinically significant gastric emptying abnormality
* Have history or presence of acute or chronic pancreatitis or an elevation in serum lipase or amylase levels greater than 3 times the upper limit of normal (ULN)
* Have an abnormal blood pressure (BP), pulse rate, or both
* Have difficulty swallowing capsules

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Steady-state Area Under the Concentration Versus Time Curve (AUC) of Orforglipron (Fasted State) | Week 3 Through Week 16
  PK: Steady-state AUC of Orforglipron (Fasted State)
PK: Steady-state Maximum Concentration (Cmax) of Orforglipron (Fasted State) | Week 3 Through Week 16
  PK: Steady-state Cmax of Orforglipron (Fasted State)
PK: Steady-state AUC of Orforglipron (Fed State) | Week 3 Through Week 16
  PK: Steady-state AUC of Orforglipron (Fed State)
PK: Steady-state Cmax of Orforglipron (Fed State) | Week 3 Through Week 16
  PK: Steady-state Cmax of Orforglipron (Fed State)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Japan (3):
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - Sumida Hospital, Sumida-ku, Tokyo
  - Hakata Clinic, Fukuoka

IPD SHARING:
Plan to Share IPD: No